CLINICAL TRIAL: NCT06613594
Title: Effects of Kaltenborn Translatoric Glides As Compared to Traction Mobilization in the Management of Frozen Shoulder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/28
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-08

CONDITIONS: Adhesive Capsulitis
Keywords: chronic pain, kaltenborn traction, kaltenborn linear translatoric glides
MeSH Terms: conditions — Bursitis; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having three groups. One group will receive conventional physical therapy, the second will receive conventional physical therapy along with kaltenborn linear translatoric glides and third group recevied conventional therapy along with kaltenborn traction mobilization. All groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional Physical Therapy Group (Active Comparator): Patients in this group will recieve conventional physical therapy including Hot pack and Tens for 10 to 15 minutes.Broomstick ROM exercises such as Internal & external rotation,Extension,flexion,abduction,these are Low intensity, short duration, 1-5 sec, 2-3 times/day, pain free passive, 3 sets of 10 reps with 1 minute rest in between will be given, Codman circular motion exercises(1time clockwise ,1 time anticlcock wise) 2-3 times/day with 10reps .Strengthening exercises include Isometric in all planes, 5 second holds, 1 set of 10 each direction, against wall.Every session will be given for 30 minutes and a total of 10 sessions would be conducted over a period of 2 weeks.
  Interventions: Other: Conventional physical therapy
- Conventional physical therapy+kaltenborn traction Group (Experimental): Patients will recieve kaltenborn traction mobiliztion in addition to conventional physical therapy including Hot pack and tens for 10 to 15 minutes , Broomstick ROM exercises such as Flexion, Internal & external rotation,Extension, Abduction,these are Low intensity, short duration, 1-5 sec, 2-3 times/day with 10 reps, pain free passive, AAROM.Codman circular motion exercises (1time clockwise ,1 time anticlockwise) 2-3 times/day with 10 reps. kaltenborn direction non specific traction mobilization for (1 minute), 3 sets of 10 reps with 1 minute rest in between will be given. Strengthening exercises include Isometric in all planes, 5 second holds, 1 set of 10 each direction, against wall.Every session will be given for 30 minutes and a total of 10 sessions would be conducted over a period of 2 consecutive weeks.
  Interventions: Other: Conventional physical therapy; Other: Kaltenborn traction mobilization
- Conventional physical therapy+kaltenborn translatoric glides Group (Experimental): Patient will recieve kaltnborn linear translatoric glides in addittion to Conventional physical therpay including Hot packs and tens for 10-15 minutes. Broomstick ROM exercises such as flexion,Exention,Internal rotation,External roation and Abuction,these are low intensity,short duration,1- 5sec,2-3 times/ day with10 reps,pain free passive, AAROM.Codman exercises circular motion exercises (1time clock wise ,1Time anticlockwise), 2-3 times/day with 10reps. Kaltenborn direction specific linear tranlatoric glides, rhtymic 5reps of each glide,such anterior glide for extension and external rotation,caudal glide for abduction,post glide for flexion and internal roation,these3 sets of painless glides will perfromed with 10 reps,rest of 1 minutes between these sets. Strengthening exercises including Isometric in all planes,5sec hold,1 sets of 10 each direction against wall. Every session will be given for 30 minutes and a total of 10 session would be conduted over a period of 2 weeks.
  Interventions: Other: Conventional physical therapy; Other: Kaltenborn translatoric glides

INTERVENTIONS:
Other: Conventional physical therapy — Patients will receive hot pack, Broom stick ROM exercises, Codman and strengthening exercises. A total of 10 sessions, 5 sessions per week for 2 consecutive weeks.
Other: Kaltenborn traction mobilization — kaltenborn direction non specific traction mobilization for (1 minute), 3 sets of 10 reps with 1 minute rest in between will be given.
  Arms: Conventional physical therapy+kaltenborn traction Group
Other: Kaltenborn translatoric glides — Kaltenborn direction specific linear tranlatoric glides, rhtymic 5reps of each glide, such anterior glide for extension and external rotation, caudal glide for abduction,post glide for flexion and internal roation,these3 sets of painless glides will performed with 10 reps,rest of 1 minutes between these sets.
  Arms: Conventional physical therapy+kaltenborn translatoric glides Group

SUMMARY:
Frozen shoulder is a common musculoskeletal condition. Painful gradual loss of both active and passive gleno-humeral motion resulting from progressive fibrosis and ultimate contracture of the gleno-humeral joint capsule.Range of motions and capsular pattern affected in frozen shoulder. Physiotherapists have a wide range of options in managing frozen shoulder including Electrotherapeutic modalities, kaltenborn mobilization, Maitland's mobilization,Mulligan's mobilization and Manipulation. So far studies have shown the efficacy of different treatments in combination or in isolation.some studies on Kaltenborn mobilization , but no obseved comparative effects of Kaltenborn mobilization i.e translatoric glides and traction mobilzation in patients with frozen shoulder.In clinically both techniques of kaltenborn are used but there is no evidence regarding which one is more effective. .If found effective,this study can help to use best clinical treatment in the managemnent of frozen shoulder.

DETAILED DESCRIPTION:
Frozen shoulder is a common MSK condition with an insidious onset accompanied by stiffness and trouble sleeping on the affected side.This condition effects General population 2-5% globally, diabetics 10-20%. Women have a significantly higher incidence males 70% of cases are female.frozen shoulder is a painful, gradual loss of both active and passive gleno-humeral motion resulting from progressive fibrosis and ultimate contracture of the gleno-humeral joint capsule.

The capsule in frozen shoulder tightens,thickness and adheres to bone it causes severe limiting of both osteikinetics and arthrokinetics shoulder range of motion,resulting in long term functional disability.As the capsule thickens mobility limitations occurs in capsular pattern.Kalternborn traction mobilization helpful in breaking capsular adhesions and decreasein severe pain, Improving shoulder limitation such as external roation ,abduction and internal rotation kaltnborn translatoric glides effective.

These mobilization changes the relative capsular adhesions and reduce stress on Gleno-humeral joint.

In clinically both techniques of kaltnborn joint mobilization are used but there is no evidence which one is more effective in the management of frozen shoulder.

Hence the current study will investigate the effects of Kaltenborn linear tranlatoric glides as compared to traction mobilization mobilization on shoulder range of motion and pain in patients with adhesive capsulitis.

This study includes Subjects with nonspecific adhesive capsulitis without specific identifiable etiology (i.e. infection, inflammatory disease) ,40-65 years of age both males and females and chronic shoulder pain > 3 months,positive capsular pattern.The selection of subjects will be using non-probability purposive sampling technique.Participants will be randomized using sealed envelope method and allocated to one of the 3 groups.

The data collection tools for pain is VAS, for ROM goniometer is used , for FEAR used fear avoidance belief questionnaire and for functional disablity is SPADI.

The time duration for treatment protocol is total of 10 sessions, 5 sessions per week for 2 consecutive weeks for approximately 25-30 mins.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Nonspecific frozen shoulder without specific identifiable etiology (i.e. infection, inflammatory disease)
* 40-65 years of age both males and females.
* Chronic shoulder pain > 3 months.
* Positive capsular pattern.

Exclusion Criteria:

* Patients with other shoulder joint pathologies, such as fractures or dislocations, glenohumeral instability or rotator cuff pathologies in the affected shoulder.
* Subjects who have undergone surgery or have experienced an acute trauma to the shoulder.
* Individuals with current or history of neurological disorders (such as stroke, Alzheimer's, or Parkinson's), rheumatologic diseases (such as rheumatoid arthritis or systemic lupus erythematous), or systemic illnesses (such as thyroid disease).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Fear Avoidance belief | 2 weeks
  fear of pain to do movement will be assessed by using fear avoidance belief questionnaire .
Pain Intensity | 2 weeks
  Pain will be assessed using Visual Analog scale which is 0-100 item scale.

SECONDARY OUTCOMES:
Shoulder Range of motion | 2 weeks
  Range of motion will be assessed using universal goniometer.
Shoulder Disability | 2 weeks
  Shoulder Disability will be assessed using shoulder pain and disability index.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan